CLINICAL TRIAL: NCT00755898
Title: Urinary Excretion of Acetylamantadine by Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); BioMark Technologies Inc. (Industry)
Responsible Party: Principal Investigator, DanielSitar, Professor Emeritus, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B2003:089
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: cancer; diagnostic test; urine; amantadine acetylation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients with a medical diagnosis of cancer appearing at outpatient clinics for treatment and/or monitoring of their disease status
  Interventions: Drug: Ingestion of a 200 mg dose of amantadine hydrochloride
- 2 (Active Comparator): Healthy adult volunteers
  Interventions: Drug: Ingestion of a 200 mg dose of amantadine hydrochloride

INTERVENTIONS:
Drug: Ingestion of a 200 mg dose of amantadine hydrochloride — Volunteer cancer patients ingest 2 x 100 mg tablets of amantadine hydrochloride with a glass of cold water 2 hours after supper.
  Arms: 1
Drug: Ingestion of a 200 mg dose of amantadine hydrochloride — Healthy subject ingests 2 x 100 mg tablets of amantadine hydrochloride with a glass of cold water 2 hours after supper
  Arms: 2

SUMMARY:
The investigators have determined that the drug amantadine hydrochloride is metabolized by acetylation by a specific enzyme named spermidine/spermine N-acetyltransferase (SSAT). This enzyme is increased in cancer cells. The investigators hypothesized that the amount of N-acetylamantadine excreted in urine during the first 12 hours after an oral dose would serve as a diagnostic biomarker for the presence of cancer in a human test subject.

DETAILED DESCRIPTION:
When patients present to their physician with symptoms of cancer at a later stage of development, survival tends to be poorer. Earlier diagnosis of cancer is expected to provide improved survival of patients due to earlier treatment intervention. However, implementation of this screening process is impaired by access and by cost. A simple and inexpensive test would serve as a screening tool that could be safely repeated at regular intervals to identify persons for whom more expensive and less accessible diagnostic investigations might become more appropriately directed. The specificity for an enzyme that increases markedly in cancer tissue, and the ease of administration of an already licensed pharmaceutical prescription product, amantadine hydrochloride, would appear to provide promise of such a desirable screening test.

ELIGIBILITY:
Inclusion Criteria:

* Either a medical diagnosis of cancer, or determination of general good health after a medical check-up within two weeks of participation in the study

Exclusion Criteria:

* Allergy to amantadine hydrochloride
* Chronic liver or kidney disease
* Chronic disease state not controlled by drug therapy, e.g. hypertension
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-12; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Amount of N-acetylamantadine excreted in a 12 hour urine sample collected after a single oral dose of amantadine hydrochloride ingested two hours after supper | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Sitar, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Bras AP, Janne J, Porter CW, Sitar DS. Spermidine/spermine n(1)-acetyltransferase catalyzes amantadine acetylation. Drug Metab Dispos. 2001 May;29(5):676-80. PMID 11302933
- [Background] Bras AP, Hoff HR, Aoki FY, Sitar DS. Amantadine acetylation may be effected by acetyltransferases other than NAT1 or NAT2. Can J Physiol Pharmacol. 1998 Jul-Aug;76(7-8):701-6. doi: 10.1139/cjpp-76-7-8-701. PMID 10030449